CLINICAL TRIAL: NCT02799615
Title: Multicenter Non-Therapeutic Study of Infliximab for Severe Refractory Colitis in Hospitalized Children
Brief Title: Anti-TNF Therapy for Refractory Colitis in Hospitalized Children
Acronym: ARCH
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0063; 2015-8753
Record Dates: First submitted 2016-06-09; First posted 2016-06-15 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2019-07

CONDITIONS: Colitis, Ulcerative; Bowel Diseases, Inflammatory
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, blood DNA, serum, plasma, colon endoscopic biopsy tissue (RNA/DNA/Formalin-fixed), stool (DNA and supernatant)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab — No standard dosing regimen will be used and the dose of infliximab will be determined by the treating physician
  Other Names: Remicade

SUMMARY:
This multicenter study is being conducted to determine whether infliximab exposure after an initial infusion is predictive of early clinical response in hospitalized pediatric patients with severe steroid-refractory UC or IBD-U. This pilot and feasibility study will establish the infrastructure, demonstrate feasibility, and collect preliminary data to support the full study.

DETAILED DESCRIPTION:
This is a multicenter prospective non-interventional cohort study to identify clinical and biological markers that predict non-response in hospitalized pediatric patients with severe corticosteroid-refractory UC or inflammatory bowel disease unspecified (IBD-U) being initiated on infliximab.

Patients hospitalized with severe UC or IBD-U (PUCAI ≥ 65 on admission) and failing intravenous corticosteroids will be eligible. Blood, stool, and rectal biopsies (if sigmoidoscopy performed for clinical indications) will be collected for translational studies (Aim 3). Patients will receive infliximab per the dose and regimen determined by clinical physician. No standard dosing regimen will be used and the dose of IFX will be determined by the treating physician. Serial PUCAI scores and infliximab levels will be obtained.

Those who are eligible to participate will have serial blood samples taken in association with drug infusions to perform pharmacokinetic/pharmacodynamic modeling of infliximab exposure. Clinical response will be determined using the Pediatric UC Activity Index (PUCAI) questionnaire.

Initially, 6 centers will participate with a minimum target enrollment goal of 36 evaluable pediatric research participants (to a maximum of 40) age > 4 years or < 18 years old with UC or IBD-U (average 6/center).

The primary endpoint will be the relationship between IFX exposure (area under the curve of the PK model) and Day 7 clinical response defined as Pediatric Ulcerative Colitis Activity Index (PUCAI) ≤ 35. Secondary endpoints will be Week 8 clinical remission, and Week 26 steroid-free, colectomy-free remission. We will initially enlist 6 centers, and enroll 36-40 evaluable patients in 2 years.

This study described by this protocol is designed as pilot and feasibility study, which we anticipate will ultimately be expanded to larger study. Therefore, to demonstrate feasibility and begin the development of a biorepository on this patient population, certain biospecimens will be collected for this study and anticipated future translational studies as follows:

* Blood will be used for IFX pharmacokinetic assays (e.g. levels, antibodies) and future biomarker discovery.
* Blood DNA we anticipate will be used for genotype/phenotype correlations and genetic predictors of rapid infliximab clearance and non-response.
* Colon tissue RNA will be used for determining how local gene expression patterns predict or explain infliximab clearance or non-response.
* Colon tissue DNA we anticipate will be used for studies of how the microbiome or epigenetic changes relate to severe UC or response to infliximab.
* Colon tissue will be used for determining the relationship between tissue TNF levels (or other proteins) and infliximab clearance or non-response.
* Stool will be collected for serial measurement of fecal calprotectin and future microbiome studies

ELIGIBILITY:
Inclusion Criteria:

1. Age criteria: ≥ 4 or < 18 years of age
2. Diagnosis of UC or IBD-U by established criteria
3. Admitted to the hospital
4. Colitis extending beyond the rectosigmoid colon
5. PUCAI ≥ 65 at admission and ≥ 45 at first dose of infliximab
6. Treatment with infliximab considered by the treating physician
7. Anticipated follow-up ≥ 6 months from infliximab initiation
8. Permission/assent of parent/guardian and research participant.

Exclusion Criteria:

1. Diagnosis of Crohn's disease
2. Enteric infection with a bacterial pathogen (including clostridium difficile), per review of medical records
3. Colon tissue positive for CMV by PCR, immunohistochemistry, or in situ hybridization, per review of the medical records
4. Colitis currently extending only to the rectosigmoid colon (proctosigmoiditis)
5. Prior treatment with infliximab or other anti-TNF agent
6. Prior treatment with cyclosporine or tacrolimus
7. PUCAI < 45 the day of first infliximab infusion
8. Pregnancy, per review of medical records and verbal report
9. Other poorly controlled medical condition
10. Hepatic disease (AST or Alk Phos > 3 times the upper limit of normal) in the absence of IBD associated liver disease
11. Renal disease (BUN and creatinine >1.5 times the upper limit of normal)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Research participants age 4 to 17 will be eligible for this study. Our target is a minimum of 36 evaluable research participants (to a maximum of 40) across up to 6 participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-05; Primary Completion 2019-02-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the relationship between IFX exposure (area under the curve of the PK model) and Day 7 clinical response defined as Pediatric Ulcerative Colitis Activity Index (PUCAI) <35. | 7 days
  IFX exposure and Day 7 PUCAI

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, MD, MSCI, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (7):
- United States (6):
  - Connecticut Children's Hospital Medical Center, Hartford, Connecticut
  - Emory University School of Medicine, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whaley KG, Xiong Y, Karns R, Hyams JS, Kugathasan S, Boyle BM, Walters TD, Kelsen J, LeLeiko N, Shapiro J, Waddell A, Fox S, Bezold R, Bruns S, Widing R, Haberman Y, Collins MH, Mizuno T, Minar P, D'Haens GR, Denson LA, Vinks AA, Rosen MJ. Multicenter Cohort Study of Infliximab Pharmacokinetics and Therapy Response in Pediatric Acute Severe Ulcerative Colitis. Clin Gastroenterol Hepatol. 2023 May;21(5):1338-1347. doi: 10.1016/j.cgh.2022.08.016. Epub 2022 Aug 27. PMID 36031093